CLINICAL TRIAL: NCT01724697
Title: Safety and Efficacy of Human Autologous Bone Marrow Stem Cells for Treatment of HBV-related Liver Cirrhosis
Brief Title: Safety and Efficacy of Human Bone Marrow Stem Cells for Treatment of HBV-related Liver Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Chinese Academy of Medical Sciences (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Han Ying, professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120912-1
Record Dates: First submitted 2012-10-31; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Liver Cirrhosis; End Stage Liver Disease
Keywords: liver cirrhosis; end stage liver disease; HBV; autologous; stem cell; bone morrow
MeSH Terms: conditions — Liver Cirrhosis; End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional treatment (Active Comparator): conventional treatment & antivrial treatment.
  Interventions: Other: conventional treatment & antivrial treatment
- BMSC transplantation (Experimental): conventional treatment & antiviral treatment & autologous bone marrow stem cell transplantation via hepatic artery
  Interventions: Other: BMSC transplantation

INTERVENTIONS:
Other: BMSC transplantation — Patients randomized to the intervention arm will be collected for bone marrow stem cells and then infused with these cells via hepatic artery.
  Arms: BMSC transplantation
Other: conventional treatment & antivrial treatment — Participants will recieve conventional treatment and antivrial treatment.
  Arms: conventional treatment

SUMMARY:
HBV related Liver disease is a common medical problem in China. An estimated 7.18% of the Chinese (about 93 million) is infected with hepatitis B, and most of the HBV- related hepatitis can developed into liver cirrhosis.

Liver transplantation is the only available life saving treatment for patients with end stage liver disease. However, lack of donors, surgical complications, rejection, and high cost are serious problems.

stem cells(SCs) possess plasticity and have the potential to differentiate into hepatocyte; Thus, SCs hold great hope for therapeutic applications. Adult bone marrow is the most common source of SCs for clinical applications.Previous study showed that bone marrow derived stem cells (BMSCs) replace hepatocytes in injured liver, and effectively rescue experimental liver failure and contribute to liver regeneration. In this study, the patients with HBV-related liver cirrhosis will undergo administration of human autologous BMSCs via hepatic artery to evaluate the safty and efficacy of human autologous BMSCs treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. HBV-related liver cirrhosis
3. Child-Pugh score 9-15
4. Written consent

Exclusion Criteria:

1. Hepatocellular carcinoma or other malignancies
2. Severe problems in other vital organs(e.g.theheart,renal or lungs)
3. Pregnant or lactating women
4. Severe bacteria infection
5. Anticipated with difficulty of follow-up observation
6. Other candidates who are judged to be not applicable to this study by doctors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
one year survival rate | one year after treatment

SECONDARY OUTCOMES:
MELD score | 1week, 4weeks, 3months, 6months, 9 months and 1year after treatment
AFP | 1week, 4weeks, 3months, 6months, 9 months and 1year after treatment
renal function | 1week, 4weeks, 3months, 6months, 9 months and 1year after treatment
child score | 1week, 4weeks, 3months, 6months, 9 months and 1year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daiming Fan, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital of Digestive Disease, Xi'an, Shaanxi, China